CLINICAL TRIAL: NCT05743270
Title: A Phase 2, Open-label, Multicenter Study Investigating Oncolytic Immunotherapy in Combination With Other Therapy in Patients With Locoregionally Advanced or Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of RP3 in Combination With Nivolumab and Other Therapy in Patients With Locoregionally Advanced or Recurrent SCCHN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Replimune Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP3-002
Record Dates: First submitted 2023-02-08; First posted 2023-02-24 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Locally Advanced Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma
Keywords: Squamous cell carcinomas of head and neck; Immunotherapy; Immuno-oncology; Oncolytic virus; Oncolytic immuno-gene therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Paclitaxel; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LA Cohort: RP3 in combination with CCRT followed by nivolumab in Locally Advanced SCCHN (Experimental): RP3 will be administered via direct intratumoral injection or via CT, ultrasound, or laryngoscopy guided intratumoral injection into superficial, subcutaneous (SC), or nodal lesions and into deeper lesions, including visceral lesions.
  Interventions: Biological: RP3; Other: CCRT(concurrent chemoradiation therapy); Biological: nivolumab
- LA Cohort: concurrent chemoradiation therapy in Patients With Locoregionally Advanced SCCHN (Active Comparator): standard-of-care CCRT (defined as intensity-modulated radiation therapy [IMRT] and cisplatin
  Interventions: Other: CCRT(concurrent chemoradiation therapy)
- R/M Cohort:RP3 in combination with carboplatin, paclitaxel and then nivolumab in R/M SCCHN (Experimental): RP3 will be administered via direct intratumoral injection or via CT, ultrasound, or laryngoscopy guided intratumoral injection into superficial, subcutaneous (SC), or nodal lesions and into deeper lesions, including visceral lesions.
  Interventions: Biological: RP3; Other: carboplatin and paclitaxel; Biological: nivolumab

INTERVENTIONS:
Biological: RP3 — Genetically modified herpes simplex type 1 virus
  Arms: LA Cohort: RP3 in combination with CCRT followed by nivolumab in Locally Advanced SCCHN; R/M Cohort:RP3 in combination with carboplatin, paclitaxel and then nivolumab in R/M SCCHN
Other: CCRT(concurrent chemoradiation therapy) — CCRT consisting of intensity modulated radiation therapy combined with a cis-platinum
  Arms: LA Cohort: RP3 in combination with CCRT followed by nivolumab in Locally Advanced SCCHN; LA Cohort: concurrent chemoradiation therapy in Patients With Locoregionally Advanced SCCHN
Other: carboplatin and paclitaxel — chemotherapeutic agents
  Arms: R/M Cohort:RP3 in combination with carboplatin, paclitaxel and then nivolumab in R/M SCCHN
Biological: nivolumab — anti-PD1 monoclonal antibody
  Arms: LA Cohort: RP3 in combination with CCRT followed by nivolumab in Locally Advanced SCCHN; R/M Cohort:RP3 in combination with carboplatin, paclitaxel and then nivolumab in R/M SCCHN

SUMMARY:
This is a Phase 2, multicenter, open-label, 2-cohort (Locoregionally Advanced Cohort or Recurrent/Metastatic Cohort) study evaluating RP3 in combination with concurrent chemoradiation therapy (CCRT) followed by nivolumab (for the LA Cohort) or combined with chemotherapy and nivolumab (for the R/M Cohort) in patients with advanced, inoperable squamous cell carcinomas of the head and neck (SCCHN), including of the oral cavity, oropharynx, hypopharynx, larynx, or unknown primary.

DETAILED DESCRIPTION:
RP3 is a genetically modified herpes simplex type 1 virus (HSV-1) that expresses exogenous genes (anti-CTLA-4 antibody, CD40 ligand and h4-1BBL) designed to directly kill tumor cells and generate a systemic anti-tumor immune response

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx or of a lymph node(s) anywhere in levels I to V of the neck that has been excluded clinically from association with cancer from a non-head and neck site
* All patients Must be willing to consent to provide archival or fresh tumor biopsy samples obtained within 60 days prior to initiation of study treatment. Patients must also consent to provide on-treatment biopsies as per protocol.
* At least 1 measurable lesion of ≥ 1 cm in longest diameter (or shortest diameter for lymph nodes), in accordance with RECIST.
* At least injectable tumors of at least 1 cm in aggregate overall longest diameter.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 -1.

Locally Advanced Cohort Only

• patients must not be amenable to surgery with curative intent

Previously untreated high-risk disease meeting at least 1 of the following criteria:

* Oral cavity, hypopharynx, larynx, oropharynx (p16 negative): Stage III/ IV Note: Cancers of the oral cavity, hypopharynx, and larynx are eligible irrespective of p16 status. These patients will not be stratified by p16 status.
* For p16 positive oropharynx cancers, patients must have either

  * T3 and/or N2 or greater disease with active smoking and/or greater than 20 pack year smoking history OR
  * T4 and/or N3 disease irrespective of tobacco use
* SCCHN of unknown primary Stage III/IV irrespective of p16 status or smoking status.
* Eligible for definitive CCRT with curative intent.

R/M Cohort Only

* Has recurrent or metastatic SCCHN eligible for first line systemic therapy for R/M disease.
* Has a PD-L1 CPS <20.

Exclusion Criteria:

* Primary tumors of nasopharynx, paranasal sinuses, nasal passages, salivary gland, thyroid or parathyroid gland, or skin.
* Tumors with histopathology indicating the tumor has sarcomatous, sarcomatoid, verrucous, mixed, undifferentiated, or otherwise nonsquamous components.
* Has an airway that is not deemed safe and stable on flexible fiberoptic laryngoscopy (FFL) performed by a head & neck cancer specialist within 7 days of first RP3 injection.
* Has a baseline serum albumin (at Screening) <2.5 g/dL and/or evidence of cachexia or muscle wasting during physical exam at Screening.
* Known acute or chronic hepatitis B or acute or chronic hepatitis C
* Systemic infection requiring intravenous (IV) antibiotics
* Active significant herpetic infections or prior complications of HSV-1 infection (eg, herpetic keratitis or encephalitis)
* History of interstitial lung disease.
* History of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
* Patients who require intermittent or chronic use of systemic (oral or IV) antivirals with known antiherpetic activity (eg, acyclovir).
* Administration of live vaccine within 28 days prior to the first dose of study treatment.
* History of allergy or sensitivity to study drug components or prior monoclonal antibody treatment.
* History of life-threatening toxicity related to prior immune treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* History of viral infections according to the protocol
* Treatment with botanical preparations within 2 weeks prior to treatment.
* Major surgery ≤ 2 weeks prior to starting study treatment.

LA Cohort only

* Has received prior radiotherapy for SCCHN.
* Has received any prior systemic therapy for SCCHN.

R/M cohort only

* Is eligible for radiation and/or surgery with curative intent.
* Has received systemic therapy for recurrence or new (ie, not present at the time of initial diagnosis) metastases of SCCHN.
* Received a paclitaxel-containing regimen as part of frontline treatment (prior to R/M disease) with a documented best response of stable disease (SD) or PD (patients who achieved a partial response [PR] or CR are eligible).
* Received a carboplatin-containing regimen as part of frontline treatment (prior to R/M disease) with a documented best response of SD or PD (patients who achieved PR or CR are eligible).
* Patients with known intolerance to carbo-platinum and/or paclitaxel, including hypersensitivity to Cremophor® EL (polyoxyethylated castor oil).
* Previously received multiple courses of irradiation to the same anatomic site unless such patient has nondoubly-irradiated, measurable, injectable lesions, which are the only lesions to be used as target lesions (for nodal disease, only lesions in nodal basins that have been previously irradiated just once or not irradiated at all may be injected and/or used as target lesions).

Note: Other protocol defined inclusion/exclusion criteria apply for each cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
LA Cohort: Progression-free Survival | From Day 1 to documented progression of disease (up to 3 years)
  Progression-free survival is defined as the time from the first day of study treatment to the date of progression of disease, which was subsequently confirmed, or death by any cause, whichever occurs first
R/M Cohort: Objective Response Rate | From Day 1 to documented progression of disease (up to 3 years)
  Percentage of subjects achieving objective response (complete response + partial response)

SECONDARY OUTCOMES:
LA Cohort: Progression-free Survival Rates at 6 and 12 Months | From Day 1 to documented progression of disease (up to 12 months)
  Progression-free survival is defined as the time from the first day of study treatment to the date of progression of disease, which was subsequently confirmed, or death by any cause, whichever occurs first
LA Cohort: Overall Survival Rate at 1, 2, and 3 Years | From Day 1 to date of death by any cause (up to 3 years)
  Overall survival is defined as the time from the first day of study treatment to the date of death by any cause
LA Cohort: Overall Response Rate and Metabolic Overall Response Rate | From Day 1 to documented progression of disease (up to 3 years)
  Overall Response Rate is the percentage of subjects achieving objective response (complete response + partial response) Metabolic overall response rate is the percentage of subjects achieving objective metabolic response (complete metabolic response + partial metabolic response)
LA Cohort: Complete Response Rate and Metabolic Complete Response Rate at 5-and 8-months Following of Initiation of Radiation Following of Initiation of Radiation | From Day 1 to documented progression of disease (up to 8Months Following of Initiation of Radiation)
  Complete response rate is the percentage of subjects achieving complete response
  Metabolic complete response rate is the percentage of subjects achieving metabolic complete response
LA Cohort: Proportion of Patients Achieving No-Evidence-of-Disease Status by Any Means (Including Salvage Surgery) | From Day 1 to end of study (up to 3 years)
  No-evidence-of-disease is defined as no evidence of malignancy at any site
LA Cohort: Cumulative Incidence of Locoregional Failure | From Day 1 to end of study (up to 3 years)
  Locoregional Failure is defined as tumor growth or disease infiltration or spread at the primary tumor location and/or at anatomic areas of local and/or regional disease.
LA Cohort: Cumulative Incidence of Distant Metastatic Failure | From Day 1 to end of study (up to 3 years)
  Distant metastatic failure is defined as growth of metastases or new appearance of metastases in lung, bone, liver, other distant organs, and/or distant lymph node stations.
LA Cohort: Duration of Clinical Benefit | From Day 1 to documented progression of disease (up to 3 years)
  Duration of clinical benefit is defined as the time from the first day of study treatment to last progression of disease, which was subsequently confirmed or with no further follow-up for response, or death due to any cause, whichever occurs first, for subjects who achieve complete response, partial response, or stable disease
LA Cohort: Summary of Patient-Reported Outcomes Measured by FACT-HNSI-22 | From Day 1 to 52 Weeks.
  FACT-HNSI-22 is a Functional Assessment of Cancer Therapy Head & Neck Cancer Symptom Index which consists of 22 items. Each item is scored in a 5 point Likert-type scale: 0=Not at all, 1=A little bit, 2=Some-what, 3=Quite a bit, and 4=Very much. The higher the score, the worse the patient outcome.
LA Cohort: Summary of Patient-Reported Outcomes Measured by EQ-5D-5L | From Day 1 to 52 Weeks
  EQ-5D-5L is a self-assessed, health related, quality of life questionnaire which consists of 2 pages: EQ-5D descriptive system and EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale which is numbered from 0 to 100. 0 means the worst health the patient can imagine. 100 means the best health the patient can imagine. The higher the score, the better the patient outcome.
LA Cohort: Frequency, Nature, and Severity of TEAEs and SAEs | From Screening through 60 days after last dose of RP3, or 100 days after last dose of nivolumab, or 28 days after last dose of either cisplatin, carboplatin, or paclitaxel, whichever occurs last
  Percentage of subjects with TEAEs and SAEs
R/M Cohort: Progression-free Survival | From Day 1 to documented progression of disease (up to 3 years)
  Progression-free survival is defined as the time from the first day of study treatment to the date of progression of disease, which was subsequently confirmed, or death by any cause, whichever occurs first
R/M Cohort: Progression-free Survival Rates at 6 and 12 Months | From Day 1 to documented progression of disease (up to 12 months)
  Progression-free survival is defined as the time from the first day of study treatment to the date of progression of disease, which was subsequently confirmed, or death by any cause, whichever occurs first
R/M Cohort: Overall Survival Rates at 1, 2, and 3 Years | From Day 1 to date of death by any cause (up to 3 years)
  Overall survival is defined as the time from the first day of study treatment to the date of death by any cause
R/M Cohort: Duration of Response | From Day 1 to documented progression of disease (up to 3 years)
  Duration of response is defined as the time from documented response until the date of progression of disease, which was subsequently confirmed or with no further follow-up, or death due to any cause, whichever occurs first
R/M Cohort: Duration of Clinical Benefit | From Day 1 to documented progression of disease (up to 3 years)
  Duration of clinical benefit is defined as the time from the first day of study treatment to last progression of disease, which was subsequently confirmed or with no further follow-up for response, or death due to any cause, whichever occurs first, for subjects who achieve complete response, partial response, or stable disease
R/M Cohort: Complete Response Rate | From Day 1 to documented progression of disease (up to 3 years)
  Percentage of subjects achieving a complete response
R/M Cohort: Disease Control Rate | From Day 1 to documented progression of disease (up to 3 years)
  Percentage of patients achieving complete response, partial response, or stable disease
R/M Cohort: Number of Patients Who Undergo Attempted Definitive Resection | From Day 1 to end of study (up to 3 years)
  Number of Patients Who Undergo Attempted Definitive Resection
R/M Cohort: Frequency, Nature, and Severity of TEAEs and SAEs | From Screening through 60 days after last dose of RP3, or 100 days after last dose of nivolumab, or 28 days after last dose of either cisplatin, carboplatin, or paclitaxel, whichever occurs last
  Percentage of subjects with TEAEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: David Cohan, MD/FACS, Study Director — Replimune Inc.
Locations (34):
- United States (12):
  - University of California San Diego, UCSD, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Medicine Division of Hematology-Oncology, Los Angeles, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University City Center and Abington, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, UPMC, Pittsburgh, Pennsylvania
  - Jefferson Health Abington Asplunhd Cancer Pavillion, Willow Grove, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Washington / Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Czechia (3):
  - University Hospital Olomouc, Olomouc
  - FN Kralovske Vinohrady, Prague
  - Fakultni Thomayerova Nemocnice, Prague
- France (5):
  - Centre Georges Francois Leclerc, Department of Oncology, Dijon
  - Centre Leon Berard, Lyon
  - Assistance Publique Hopitaux De Marseille, Marseille
  - CHU Nimes, Instiut de Cancerologie du Gard, Medical Oncology, Nîmes
  - Institut Gustave Roussy Paris, Villejuif
- Germany (5):
  - Charite University Hospital of Berlin, Comprehensive Cancer Center, Berlin
  - Universitatsklinik Jena Klinik und Poliklinik fur Hals-, Nasen - und Ohrenheilkunde, Jena
  - University Hospital Leipzig Clinic and Polyclinic for otorhinolaryngology, Leipzig
  - LMU Klinikum, Medizinische Klinik und Poliklinikum III, Munich
  - Universitatsklinikum Ulm, Ulm
- Greece (2):
  - University General Hospital Attikon, Chaïdári
  - Agios Lukas Hospital, Thessaloniki
- Szpital Specjalistyczny im Ludwika Rydygiera w Krakowie sp z oo, Department of Clinical Oncology, Krakow, Poland
- Spain (5):
  - Vall d'Hebron University Hospital, Vall d' Hebron Institute of Oncology (VHIO), Barcelona
  - La Paz Univeristy Hospital, Universidad Autonoma de Madrid, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Fundacion Instituto Valenciano de Oncologia, Valencia
- The Royal Marsden NHS Foundation Trust, London, United Kingdom